CLINICAL TRIAL: NCT00260637
Title: A Double Blind, Sham Controlled Trial Evaluating the Efficacy of Acupuncture in Relieving Symptoms of Chronic Prostatitis/ Chronic Pelvic Pain Syndrome
Brief Title: Efficacy Study of Acupuncture to Relieve Symptoms of Chronic Prostatitis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Collaborators: University of Washington (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACUCP
Record Dates: First submitted 2005-11-29; First posted 2005-12-01 (Estimated); Last update posted 2006-10-26 (Estimated); Status verified 2005-11

CONDITIONS: Prostatitis
Keywords: Prostatitis
MeSH Terms: conditions — Prostatitis | interventions — Acupuncture Therapy

INTERVENTIONS:
Procedure: Acupuncture

SUMMARY:
Limited evidence suggests that acupuncture may help relieve symptoms of chronic prostatitis/chronic pelvic pain syndrome. This study evaluated if acupuncture twice weekly for 10 weeks would help ameliorate symptoms of CP/CPPS.

DETAILED DESCRIPTION:
Various studies have reported that this acupuncture able to relieve symptoms of chronic prostatitis (CP)/ chronic pelvic pain syndrome (CPPS). However, controversy exists on the efficacy of this technique due to poor experimental designs and lack of placebo controls in these experiment. This study is the first randomised controlled study which will evaluate if acupuncture for 10 weeks will help improve symptoms of CP/CPPS

ELIGIBILITY:
Inclusion Criteria:

* Symptoms of discomfort or pain in the pelvic region for at least a three (3) months period within the last six (6) months.
* Moderate overall score on the NIH-CPSI (overall score more than 15 out of a potential of 0-43 points)
* Diagnosed as having CPPS Category III
* Participant is willing to undergo 10 weeks of acupuncture treatment

Exclusion Criteria:

* History of prostate, bladder or urethral cancer.
* Inflammatory bowel disease (such as Crohn's disease or ulcerative colitis, but not irritable bowel syndrome).
* Undergone pelvic radiation or systemic chemotherapy, intravesical chemotherapy or intravesical BCG.
* Treated for unilateral orchialgia without pelvic symptoms.
* Active urethral stricture.
* Undergone TURP, TUIP, TUIBN, TUMT, TUNA, balloon dilation of the prostate, open prostatectomy or any other prostate surgery or treatment such as cryotherapy or thermal therapy.
* Neurological impairment or psychiatric disorder preventing his understanding of consent and his ability to comply with the protocol.
* Liver disease.
* Diagnosed as acute or chronic bacterial prostatitis.
* History of urinary tract infection positive uropathogen for the past year.
* Taking medications which could affect the lower urinary tract function
* History of type 1 or 2 diabetes.
* Treated/currently undergoing treatment with acupuncture for any other illness including prostatitis for the past 6 months.
* Refusal to be needled or any form of bleeding disorder.

Ages: 20 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86
Dates: Start 2004-02; Study Completion 2005-08

PRIMARY OUTCOMES:
Six point drop in NIH-CPSI total Score

SECONDARY OUTCOMES:
Individual domains of the NIH-CPSI
Patient reported Global Response Assessment
International Prostate Symptom Score
International Index of Erectile Function
Brief Pain Inventory- Short Form

CONTACTS AND LOCATIONS:
Overall Officials: Men L Liong, MD, Principal Investigator — Consultant Urologist; John N Krieger, MD, Principal Investigator — University of Washington; Kah H Yuen, PhD, Principal Investigator — Universiti Sains Malaysia
Locations (4):
- Malaysia (4):
  - Metro Hospital, Sungai Petani, Kedah
  - Hospital Lam Wah Ee, Batu Lanchang, Pulau Pinang
  - Hospital Pantai Mutiara, Bayan Lepas, Pulau Pinang
  - Island Hospital, George Town, Pulau Pinang

REFERENCES:
- [Derived] Lee SW, Liong ML, Yuen KH, Krieger JN. Acupuncture and immune function in chronic prostatitis/chronic pelvic pain syndrome: a randomized, controlled study. Complement Ther Med. 2014 Dec;22(6):965-9. doi: 10.1016/j.ctim.2014.10.010. Epub 2014 Oct 23. PMID 25453515
- [Derived] Lee SW, Liong ML, Yuen KH, Leong WS, Khan NK, Krieger JN. Validation of a sham acupuncture procedure in a randomised, controlled clinical trial of chronic pelvic pain treatment. Acupunct Med. 2011 Mar;29(1):40-6. doi: 10.1136/aim.2010.003137. Epub 2011 Jan 18. PMID 21245238